CLINICAL TRIAL: NCT07261722
Title: Harnessing the Power of Military Peers to Reduce Sexual Violence and Risky Drinking in Service Members
Brief Title: Collaborative Opportunities for Reducing Alcohol and Sexual Violence Together
Acronym: COAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Jennifer Read, SUNY Distinguished Professor and Chair of Department of Psychology, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 00006595; TP210286 (Other Grant/Funding Number: U.S. Department Of Defense)
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Sexual Violence; Behavior Change; Military Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer-Based Motivational Interview (PMI) (Experimental): Will participate in the Peer-Based Motivational Interview (PMI) intervention
  Interventions: Behavioral: Peer-Based Motivational Interview

INTERVENTIONS:
Behavioral: Peer-Based Motivational Interview — The intervention will use Motivational Interviewing's (MI) collaborative conversation style for strengthening commitment to change, to motivate and prepare service members to work together to reduce Sexual Violence (SV) risk. This intervention will target ways that the peer dyad may support, encourage, and share responsibility with one another in protecting against SV. The Peer-based MI (PMI) will then use the responsibility and relationship of peers as a framework to foster collaborative efforts to increase readiness and decrease barriers to helping behavior. As part of this, the PMI will focus on the identification and implementation of skills peers can use to help one another prevent SV. PMI will include a focused discussion of the ways drinking may impede helping efforts. Moreover, the PMI will encourage service members to identify personal, specific strategies for reducing the effects of alcohol on helping.

SUMMARY:
The goal of this clinical trial is to test if a modified peer-based motivational intervention (the Military PAIRS; MPAIRS) is reasonable and practical for military contexts. The main questions it aims to answer are:

* Does it works to reduce SV?
* Does it works to reduce risky drinking? To test this, participants will answer questions about their SV history and risky drinking. Then they will be given MPAIRS. After 1 month, they will be asked about their SV history and risky drinking again.

DETAILED DESCRIPTION:
The objective of the proposed study is to adapt an innovative, peer-based motivational interview (PMI) that encourages and prepares peers to reduce sexual violence (SV) risk. Delivered to pairs of peers (dyads), the PMI will be designed to foster collaborative efforts to increase readiness for, and decrease barriers to helping behavior, and to teach and plan together for assault prevention skills. As the role of alcohol has been under-addressed in SV prevention efforts, the PMI also will explicitly attend to how intoxication may serve as a barrier to peer intervention, and strategies for overcoming this barrier. The completion of this project's aims will yield a novel intervention that capitalizes on the natural resource of military responsibility to decrease risk for sexual violence - a pervasive problem affecting a substantial portion of military service members in the U.S.

Twelve peer dyads will participate in the peer-based motivational interview (PMI). The study will compare the participants at baseline to themselves at a 1 month follow up on outcomes. The study will focus on whether effects are in the expected direction and whether the strength of effect sizes are of practical magnitude. It is expected that participants will demonstrate significant increases in readiness, and engagement in peer assault prevention behavioral skills (PAPBs), and demonstrate decreases in perceived barriers. Follow-up data will be utilized to provide a rich description of the role of alcohol in implementing PAPBs, and whether the PMI reduces the impact of alcohol use. In exploratory analyses, it will be examined whether the intervention may be associated with decreased assault risk, as well as decreased drinking.

ELIGIBILITY:
Inclusion Criteria:

* Enlisted U.S. Navy service members on active duty status
* Meet criteria for risky drinking (i.e. score of 4+ for men, 2+ for women according to the AUDIT-C)
* Have an eligible peer and the pair must socialize together at least twice a month

Exclusion Criteria:

* Individuals who endorse evidence of withdrawal (Item 6 on the AUDIT)

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Readiness to intervene | Baseline and 1 month followup
  10 item scale scored on a 5 point likert type scale with higher value indicating they are more ready to intervene on behalf of the other member of the dyad in areas of concern for abuse.
  Modeled after: Center for Evidence-Based Practices at Case Western Reserve University (2010). Readiness Ruler. Center for Evidence-Based Practices, Case Western Reserve University.
Peer -Directed Bystander Behaviors Scale for Friends | Baseline and 1 month follow up
  44 item scale. The answers provided are yes/no/"I did not perceive an opportunity to do this" for each item in 3 different contexts (Friend, Stranger, Someone in Military). Each item is a situation that the participant may have been in to help someone in the past month. The participant reports if they did that helped, didn't help, or didn't have that situation for each context.
  Banyard, V. L., Moynihan, M. M., Cares, A. C., & Warner, R. A. (2014). How do we know if it works? Defining measurable outcomes in bystander-focused violence prevention. Psychology of Violence, 4(1), 101-115.
Assault Protective Strategies | Baseline and 1 month follow up
  20 item scale. It is scored on a 4 point likert type scale with an option for "I prefer to not answer" and an option for "I did not perceive an opportunity to do this". The scale is made up of items of strategies that people do either before going out, or while they are out to reduce risk for sexual assault. The participant reports to what extent they use each strategy with a higher number meaning they use the strategy to a greater extent.
PBSS-20 Alcohol Protective Strategy | Baseline and 1 month follow up
  20 item scale. It is scored on a 6 point likert type scale. The scale is made up of items of different strategies people often use to protect against negative consequences of alcohol use. The participant reports to what extent they use each strategy with a higher number meaning they use the strategy to a greater extent.
  Treloar H, Martens MP, McCarthy DM. The Protective Behavioral Strategies Scale-20: improved content validity of the Serious Harm Reduction subscale. Psychol Assess. 2015 Mar;27(1):340-6. doi: 10.1037/pas0000071.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer P Read, Ph.D., Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo Department of Psychology, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share a de-identified data set which will include baseline demographics and readiness to intervene, peer -directed bystander behaviors, peer-based assault protective strategy use, and Alcohol Protective Strategy outcomes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available once data collection is completed and conclude 5 years after.
Access Criteria: There must be an articulation of a clear research question and analytic plan by an established investigator with the relevant credentials. The information will be shared as a digital file through email.